CLINICAL TRIAL: NCT03706287
Title: Efficacy and Safety of Anlotinib Combined With Platinum Plus Pemetrexed in T790M Mutation Negative Metastastic Non-squamous Non-small-cell Lung Cancer After Progression on First-line EGFR TKI: a Phase II, Muti-center, Single Arm Study
Brief Title: Efficacy and Safety of Anlotinib Plus Platinum Plus Pemetrexed in T790M-negative NSCLC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Juan LI, MD, Director of standard treatment department of medical oncology, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-L022
Record Dates: First submitted 2018-10-07; First posted 2018-10-15 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Lung Cancer Metastatic
Keywords: non small cell lung cancer; anlotinib; pemetrexed; T790M negative
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib + AP/PC (Experimental)
  Interventions: Drug: anlotinib 8mg + AP/PC; Drug: anlotinib 10mg + AP/PC; Drug: anlotinib 12mg + AP/PC; Drug: anlotinib + AP/PC

INTERVENTIONS:
Drug: anlotinib 8mg + AP/PC — anlotinib 8mg/d, q.d., p.o. 1-14days every 21 days Pemetrexed(A) 500mg/m2, IV, Day 1; Cisplatin(P) 25mg/m2,IV,Day 1-3 or Carboplatin(C) area under curve(AUC)=5, IV, Day 1; AP or AC will be administered every 21 days starting on Day 1.
  Other Names: Pemetrexed/Cisplatin or Pemetrexed/Carboplatin
Drug: anlotinib 10mg + AP/PC — anlotinib 10mg/d, q.d., p.o. 1-14days every 21 days Pemetrexed(A) 500mg/m2, IV, Day 1; Cisplatin(P) 25mg/m2,IV,Day 1-3 or Carboplatin(C) area under curve(AUC)=5, IV, Day 1; AP or AC will be administered every 21 days starting on Day 1.
  Other Names: Pemetrexed/Cisplatin or Pemetrexed/Carboplatin
Drug: anlotinib 12mg + AP/PC — anlotinib 12mg/d, q.d., p.o. 1-14days every 21 days Pemetrexed(A) 500mg/m2, IV, Day 1; Cisplatin(P) 25mg/m2,IV,Day 1-3 or Carboplatin(C) area under curve(AUC)=5, IV, Day 1; AP or AC will be administered every 21 days starting on Day 1.
  Other Names: Pemetrexed/Cisplatin or Pemetrexed/Carboplatin
Drug: anlotinib + AP/PC — anlotinib doses to be determined following the completion of Phase I of the study, q.d., p.o. 1-14days every 21 days Pemetrexed(A) 500mg/m2, IV, Day 1; Cisplatin(P) 25mg/m2,IV,Day 1-3 or Carboplatin(C) area under curve(AUC)=5, IV, Day 1; AP or AC will be administered every 21 days starting on Day 1.

SUMMARY:
This study is conducted to explore the safety and efficacy of anlotinib, a tyrosine kinase inhibitors of vascular endothelial growth factor receptor 2（VEGFR）、FGFR（fibroblast growth factor receptor）, platelet-derived growth factor receptor（PDGFR） and tumor cell proliferation related kinase c-Kit, combined with platinum plus pemetrexed in T790M mutation negative metastatic non-squamous non-small cell lung cancer(NSCLC) after the failure of EGFR-TKI.

DETAILED DESCRIPTION:
Anlotinib, an oral highly potent tyrosine-kinase inhibitor targeting VEGFR、PDGFR、FGFR and c-kit，has demonstrated improved survival in previously treated patients with advanced non-small-cell lung cancer(NSCLC).

In the phase Ⅲ study ALTER0303, patients who failed at least two kinds of systemic chemotherapy (third line or beyond) or drug intolerance were treated with anlotinib or placebo, the anlotinib group PFS and OS were 5.37 months and 9.63 months, the placebo group PFS and OS were 1.4 months and 6.3 months. Therefore,we envisage using anlotinib plus platinum plus pemetrexed treat the EGFR wild-type metastatic non-small cell lung cancer patients who were failure in the treatment of chemotherapy with platinum containing drugs, to further improve the patient's PFS.

The study is divided into two stages，phase I use a dose escalation trial design to explore the safety, tolerability, dose-limiting toxicities(DLT), Maximum Tolerable Dose(MTD), A cohort of 3~6 subjects will be enrolled at each dose level, If 0 of 3 or ≤ 1 of 6 subjects experience a DLT, the phase I trial will move ahead to the next dose until ≥ 2 of 6 subjects experience a DLT，and the current dose will be considered the MTD. Following completion of the dose escalation trial and determination of MTD（Phase I）, a single arm study including 44 subjects may be enrolled to further evaluate safety, tolerability, and efficacy of anlotinib in combination with platinum plus pemetrexed in the same target population（phase II）. Phase II is to designed to explore the anti-tumor activity of anlotinib combined with platinum plus pemetrexed in T790M mutation negative metastatic non-squamous non-small cell lung cancer(NSCLC) after the failure of EGFR-TKI.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ 75 years of age. Signed the informed consent form prior to patient entry
* Histologically or pathologically confirmed non-squamous non-small cell lung cancer(NSCLC) with stage IV .
* Epidermal Growth Factor Receptor(EGFR)mutations confirmed by molecular detection (including, but not limited to 19 exon deletion and L858R) external pathological examination was accepted (including pathological or blood test results)
* Patients have only be treated with EGFR -TKIs（Tyrosine kinase inhibitors）including gefitinib, elotinib or icotinib, and received a best response of PR for ≥4months or SD for 6 months; disease has progressed recently according to RECIST 1.1 and negative for T790M detection（detection methods including ddPCR、ARMS or NGS） (For recurrent patients, adjuvant chemotherapy, neoadjuvant chemotherapy or neoadjuvant chemotherapy plus adjuvant were assessed for eligibility, and the last treatment time must be more than 6 months before enrollment）
* Must have at least one measurable lesion as per RECIST 1.1 defined as a lesion that is 10mm in longest diameter imaged by CT scan or MRI；prior topical treatment, such as radiotherapy cryosurgery to the lesions is not allowed in less than 3 months;
* Life expectancy ≥3 months.
* Eastern Cooperative Oncology Group(ECOG) performance status 0 or 1.
* Toxicity caused by prior anti-cancer treatments was restored to ≤ level 1 in CTC AE (4.0) , except alopecia;
* The blood routine examination need to be standard (no blood transfusion and blood products within 14 days, no g-csf and other hematopoietic stimulating factor correction) Hemoglobin（HB）≥90 g/L A Neutrophil count of （ANC）≥1.5×109/L A Platelet count of （PLT）≥80×109/L A Total bilirubin (TBil) of ≤1.5 upper normal limitation (UNL) A alanine aminotransferase (ALT) and a aspartate aminotransferase (AST) of ≤2.5 UNL, in case of liver metastasis ALAT and ASAT≤5 UNL A creatinine (Cr) of ≤1.5 UNL; a creatinine clearance rate ≥ 60ml/min (Cockcroft-Gault)
* The woman patients of childbearing age who must agree to take contraceptive methods during the research and within another 8 weeks after it and examined as negative in blood serum test or urine pregnancy test within 7 days before the research; the man patients who must agree to take contraceptive methods during the research and within another 8 weeks;
* Voluntarily joined the study and signed informed consent, with good compliance and follow-up.

Exclusion Criteria:

* Small Cell Lung Cancer mixed or squamous mixed;
* No squamous NSCLC with hemoptysis (>50ml/day);
* Symptomatic brain metastases after treatment;
* Tumor locate within a distance of less than 5 mm from the large vessels, less than 2 cm from the bronchial tree, or has invaded local large vessels; tumor with cavum or necrotic obviously;
* Uncontrolled hypertension (systolic ≥150mmHg and/or diastolic ≥100mmHg, despite optimal drug therapy).
* Patients with with grade Ⅱ myocardial ischemia or myocardial infarction, poor control of arrhythmias (including QTc interval male ≥ 450 ms, female ≥470 ms); according to NYHA standard, grade Ⅲ ~ Ⅳ heart failure, or cardiac color Doppler ultrasound examination showed left ventricular ejection fraction (LVEF) <50%.
* Coagulation dysfunction (INR> 1.5, PT> ULN +4s or APTT> 1.5 ULN), with bleeding tendency or ongoing thrombolysis or anti-blood coagulation treatment;note: Note: under the premise of International Normalized ratio (INR) of prothrombin time (PT) Less than or equal to 1.5, allow to administrate low-dose heparin (adult daily dose is 06000 ~ 12000 U) or low-dose aspirin (100 mg daily dosage or less) , for prophylactic purposes
* Patients whose routine urine tests indicate that urine protein ≥ ++ or verifies that the 24-h urine protein quantitation ≥ 1.0 g.
* Patients whose has peripheral neuropathy over level 2 in CTC AE4.0, except trauma.
* Patients with respiratory syndrome (difficulty breathing of level 2 or higher ), serous cavity effusion need to surgical treatment ( including pleural of level 2 or higher with respiratory distress and anoxia
* Patients who have unhealed wounds or fractures for a long time.
* Patients with severe infections , and need to receive systemic antibiotic treatment
* Decompensated diabetes or other contraindication with high dose glucocorticoid therapy;
* Cirrhosis or decompensated liver disease; active or untreated hepatitis C and/or Hepatitis B virus (HBV) infection（prior hepatitis B history, HBsAg positive and HBV DNA≥500IU/mL; HCV RNA positive and hepatic Insufficiency
* History of immunodeficiency, HIV infection etc
* Active pulmonary tuberculosis;
* Has an obvious factor influencing oral drug absorption, such as unable to swallow, chronic diarrhea and intestinal obstruction, etc
* Patients who received major surgical operations or experienced severe traumatic injuries, bone fracture, or ulcers within 4 weeks before screening.
* Severe weight loss (> 10%) Within 6 weeks before Random
* Patients who had obvious hemoptysis (>50ml/day) within 3 months before screening; Patients who experienced bleeding symptoms of clinical significance within 3 months before screening, or with confirmed bleeding tendency such as hemorrhage of digestive tract, hemorrhagic gastric ulcer, baseline occult blood in stool ++ and above, or vasculitis, etc;
* Patients who manifested arterial/venous thrombus events, e.g. cerebrovascular accident (including transient ischemic attack), deep venous thrombosis and pulmonary embolism, etc., within 12 months before screening.
* Allergic reactions to anotol or excipients in experimental drugs.
* Allergic reactions to contrast medium
* Patients have participated in other antitumor drug clinical trials Within 4 weeks before enrollment or prepare to receive systemic anti-tumor treatment during the study or Within 4 weeks before randomization
* Patients with any other medical condition or reason, in that investigator's opinion, makes the patient unstable to participate in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2018-12-06 (Actual); Primary Completion 2021-03-10 (Estimated); Study Completion 2021-03-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 24 months
  PFS defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause.
Dose limiting toxicity (DLT) | Estimated about 6 months
  Dose Limiting Toxicity (DLT) is referred to grade 3 non-hematological toxicity or grade 4 hematological toxicity according to NCI CTCAE 4.03 criteria
Maximum tolerance dose (MTD) | Estimated about 6 months
  Maximum Tolerance Dose (MTD) is the dose of treatment in the cohort where there are 2 cases of DLT reported.

SECONDARY OUTCOMES:
Objective response rate(ORR) | Up to 24months
  To determine ORR of Anlotinib Anlotinib combined with Platinum-based Pemetrexed in T790M mutation negative Advanced NSCLC. ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.
Disease Control Rate (DCR) | Up to 24months
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1.
Duration of Response (DOR) | Up to 24months
  Defined as the the time from first confirmed CR or PR until the first date of either objective disease progression or death due to any cause.
Safety (Number of Participants with Adverse Events as a Measure of Safety and Tolerability) | Until 21 day safety follow-up visit
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: ping yu, Principal Investigator — Sichuan Cancer Hospital and Research Institute; juan li, doctor, Principal Investigator — Sichuan Cancer Hospital and Research Institute
Locations (6):
- China (6):
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Chengdu fifth people's hospital, Chengdu
  - People's hospital of deyang city, Deyang
  - The affiliated hospital of southwest medical university, Luzhou
  - Nanchong central hospital, Nanchong
  - Suining central hospital, Suining

IPD SHARING:
Plan to Share IPD: No